CLINICAL TRIAL: NCT06483568
Title: Behavioral Mechanisms and Health Outcomes of Positive Psychological Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Samantha J. Heintzelman, PhD, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Pro2023002402
Record Dates: First submitted 2024-04-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Well-Being, Psychological
Keywords: Emotional Well-Being; Happiness; Gratitude; Kindness; Self-Compassion; Capitalization
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to complete positive psychology intervention activities or procedure-matched activities related to personal organization.
Who Masked: Participant, Investigator
Masking Description: Participants will not be aware of whether their activities are considered the active or control activities as both will be described as self-improvement activities. The PI and all research staff interacting with participants will not be aware of their condition assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Psychology Intervention Activities (Experimental): Four week intervention with four weekly activities including gratitude journal, random acts of kindness, self-compassionate letter, and capitalizing on positive events activities.
  Interventions: Behavioral: Pathways to Happiness Intervention
- Personal Organization Activities (Sham Comparator): Control participants will complete procedure-matched activities related to personal organization, including writing in a completed tasks journal, completing a weekly task burst, productivity letter, and talking to others about tasks activities.
  Interventions: Behavioral: Personal Organization Activities

INTERVENTIONS:
Behavioral: Pathways to Happiness Intervention — Four weeks of activities including a gratitude journal, random acts of kindness, self-compassionate letter, and capitalizing on positive events activities.
  Arms: Positive Psychology Intervention Activities
Behavioral: Personal Organization Activities — Four weeks of activities including a completed tasks journal, weekly "task burst," productivity letter, and talking to others about task activities.
  Arms: Personal Organization Activities

SUMMARY:
The goal of this clinical trial is to learn if engaging in a multi-activity positive psychology intervention increases emotional well-being

The main aims of this project are to:

1. Test the efficacy of a multi-activity positive psychology intervention for increasing emotional well-being in a racial-ethnically and socioeconomically diverse sample.
2. Identify physical and social behavioral mechanisms driving positive psychology intervention effects on emotional well-being change and the durability of these effects over time.
3. Examine physical health outcomes stemming from emotional well-being gains.

Participants will:

Visit the laboratory three times to complete survey measures and physical assessments.

Complete brief survey items three times a day for 10 weeks of the study period. Engage with assigned activities weekly for four weeks of the study period.

DETAILED DESCRIPTION:
Participation will span 20 weeks around a four-week treatment phase. Assessments will involve three lab visits and experience sampling method surveys completed on participants' smart phones in response to short message service (SMS) message alerts.

Lab Visit 1 (Baseline): Participants will begin participation with an in-person lab visit held in small groups. This visit will begin with a guided informed consent procedure. Participants will complete baseline self-report measures and physiological assessments and receive procedure instructions.

Pre-Intervention Monitoring (weeks 1 & 2): For two weeks, participants will compete three very brief experience sampling surveys per day.

Random Assignment, Treatment and Monitoring (weeks 3,4,5,& 6): Participants will be randomly assigned to the online four-week Pathways to Happiness treatment condition or a matched activity control condition. All participants will complete the four weeks of activities (either Pathways to Happiness Positive Psychology Intervention (PPI) or control activities) on the Pathways to Happiness platform. They will complete weekly check-in items on the Pathways to Happiness platform to assess their compliance with the activity instructions and their experiences with the activities. Participants in both conditions will continue completing experience sampling surveys during this time.

Lab Visit 2 (Post-Test), after week 6: The second lab visit will occur after week six, following the treatment phase. It will involve identical questionnaires and physiological screenings as in the baseline visit.

Post-Intervention Monitoring (weeks 7&8): After the treatment phase, two weeks of post-intervention experience sampling survey monitoring will begin.

Waiting Period: Participants will not engage in any formal study activities from weeks 9 to 19.

Follow-Up Monitoring (weeks 19-20): Follow-up experience sampling monitoring will commence for the final two weeks of the study, 10 weeks after the previous monitoring period.

Lab Visit 3 (Follow-Up), after week 20: The final lab visit, identical to the others, will occur after week 20 and will conclude with an exit interview regarding participants' experiences in the study and with each PPI activity.

ELIGIBILITY:
Inclusion Criteria:

* Fluent or native English speaker capable of completing survey questionnaires in English

Exclusion Criteria:

* Major depressive disorder (PHQ-9 > or = 15)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Life Satisfaction | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Satisfaction with Life Scale, 1-7 scale, higher scores better
Positive Affect | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Scale of Positive and Negative Affect, 1-5 scale, higher scores better
Negative Affect | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Scale of Positive and Negative Affect, 1-5 scale, lower scores better
Meaning in Life | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Meaning in Life Questionnaire, 1-7 scale, higher scores better
Optimism | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Life Orientation Test-Revised, 1-5 scale, higher scores better
Perceived General Health | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Medical Outcomes Study (MOS) Short Form Health Survey (SF-36), General Health Perceptions Subscale, 1-5, higher scores better
Blood Pressure | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Systolic and Diastolic Blood Pressure In-lab measurement with OMRON 10 Series Wireless Upper Arm Blood Pressure Monitor
Heart Rate | baseline, immediate post-treatment, 14-week post-treatment follow-up
  In-lab measurement with OMRON 10 Series Wireless Upper Arm Blood Pressure Monitor
Peak Expiratory Flow Rate | baseline, immediate post-treatment, 14-week post-treatment follow-up
  In-lab measurement with EasyOne Air Spirometer
Grip Strength | baseline, immediate post-treatment, 14-week post-treatment follow-up
  In-lab measurement with Jamar Plus+ Digital Hand Dynamometer
Momentary Mood | 3x daily; weeks 1-8, 19, 20
  Rate your current mood. 1 (very bad) to 7 (very good), higher scores better
Momentary Meaning in Life | 3x daily; weeks 1-8, 19, 20
  Daily Meaning Scale, 1-7, higher scores better

SECONDARY OUTCOMES:
Amusement | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Dispositional Positive Emotions Scale, 1-7, higher scores better
Awe | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Dispositional Positive Emotions Scale, 1-7, higher scores better
Compassion | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Dispositional Positive Emotions Scale, 1-7, higher scores better
Contentment | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Dispositional Positive Emotions Scale, 1-7, higher scores better
Joy | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Dispositional Positive Emotions Scale, 1-7, higher scores better
Love | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Dispositional Positive Emotions Scale, 1-7, higher scores better
Pride | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Dispositional Positive Emotions Scale, 1-7, higher scores better
Hope | baseline, immediate post-treatment, 14-week post-treatment follow-up
  State Hope Scale, 1-8, higher scores better
Depression | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Patient Health Questionnaire-9, 0-27, lower scores better
Anxiety | baseline, immediate post-treatment, 14-week post-treatment follow-up
  State-Trait Anxiety Inventory, 1-4, lower scores better
Perceived Stress | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Perceived Stress Scale, 0-4, lower scores better
Loneliness | baseline, immediate post-treatment, 14-week post-treatment follow-up
  UCLA Loneliness Scale, 1-4, lower scores better
Social Connectedness | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Comprehensive Inventory of Thriving, 1-5, higher scores better
Social Support | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Perceived Social Support Scale, 1-5, higher scores better
Sleep Quality | baseline, immediate post-treatment, 14-week post-treatment follow-up
  Pittsburgh Sleep Quality Index, 0-21, lower scores better
Cigarette Use | baseline, immediate post-treatment, 14-week post-treatment follow-up
  cigarette smoking days/month x cigarettes per average smoking day, lower scores better
Tobacco Use (non-cigarette products) | baseline, immediate post-treatment, 14-week post-treatment follow-up
  tobacco use days/month x average uses per day of using, lower scores better
Alcohol Use | baseline, immediate post-treatment, 14-week post-treatment follow-up
  days in last month drinking x average number of drinks/drinking day, lower scores better
Vigorous Activity Level | baseline, immediate post-treatment, 14-week post-treatment follow-up
  International Physical Activity Questionnaire, days/week x minutes/day, higher scores better
Moderate Activity Level | baseline, immediate post-treatment, 14-week post-treatment follow-up
  International Physical Activity Questionnaire, days/week x minutes/day, higher scores better
Walking | baseline, immediate post-treatment, 14-week post-treatment follow-up
  International Physical Activity Questionnaire, days/week x minutes/day, higher scores better
Physical Functioning | baseline, immediate post-treatment, 14-week post-treatment follow-up
  MOS Short Form Health Survey (SF-36), Physical Functioning Subscale, 1-3, higher scores better
Role Functioning--Physical | baseline, immediate post-treatment, 14-week post-treatment follow-up
  MOS Short Form Health Survey (SF-36), Physical Role Functioning Subscale, 0-4, lower scores better
Role Functioning--Emotional | baseline, immediate post-treatment, 14-week post-treatment follow-up
  MOS Short Form Health Survey (SF-36), Emotional Role Functioning Subscale, 0-3, lower scores better
Social Functioning | baseline, immediate post-treatment, 14-week post-treatment follow-up
  MOS Short Form Health Survey (SF-36), Social Functioning Subscale, 0-5, lower scores better
Sitting | baseline, immediate post-treatment, 14-week post-treatment follow-up
  International Physical Activity Questionnaire, hours/weekday, lower scores better
Bodily Pain | baseline, immediate post-treatment, 14-week post-treatment follow-up
  MOS Short Form Health Survey (SF-36), Pain Subscale, 2-11, lower scores better
General Mental Health | baseline, immediate post-treatment, 14-week post-treatment follow-up
  MOS Short Form Health Survey (SF-36), General Mental Health Subscale, 1-6, higher scores better
Vitality | baseline, immediate post-treatment, 14-week post-treatment follow-up
  MOS Short Form Health Survey (SF-36), Vitality Subscale, 1-6, higher scores better
Momentary physical activity | 3x daily; weeks 1-8, 19, 20
  Physical activity behaviors checklist, 0-3, higher scores better
Momentary tobacco use | 3x daily; weeks 1-8, 19, 20
  Have you used a tobacco product in the previous 4 hours? 0 (no)/1(yes), lower scores better
Momentary alcohol use | 3x daily; weeks 1-8, 19, 20
  Have you consumed alcohol in the previous 4 hours? 0 (no)/1(yes), lower scores better
Momentary eating | 3x daily; weeks 1-8, 19, 20
  Have you eaten [fruit or vegetable/sugary dessert, snack, or beverage] in the previous 4 hours? 0-2, higher scores better
Momentary connective Behaviors | 3x daily; weeks 1-8, 19, 20
  Connective behaviors checklist, 0-5, higher scores better
Momentary Stress | 3x daily; weeks 1-8, 19, 20
  How stressed do you feel right now? 1(not at all) to 7 (very much), lower scores better
Momentary Depression | 3x daily; weeks 1-8, 19, 20
  How depressed do you feel right now? 1(not at all) to 7 (very much), lower scores better
Momentary Anxiety | 3x daily; weeks 1-8, 19, 20
  How anxious do you feel right now? 1(not at all) to 7 (very much), lower scores better
Momentary Loneliness | 3x daily; weeks 1-8, 19, 20
  How lonely do you feel right now? 1(not at all) to 7 (very much), lower scores better
Momentary Perceived General Health | 3x daily; weeks 1-8, 19, 20
  How do you feel in terms of your physical health right now? 1 (poor) to 5 (excellent), higher scores better
Sleep Quality | 1x daily; weeks 1-8, 19, 20
  How would you rate the quality of your sleep last night? 1 (very bad) to 4 (very good), higher scores better
Sleep Duration | 1x daily; weeks 1-8, 19, 20
  Wake up time - (lights out time + time to fall asleep), higher scores better
Common Symptoms Checklist | 1x daily; weeks 1-8, 19, 20
  1-5, lower scores better

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial, after deidentification, and the study protocol materials will be shared on the Open Science Framework.
Supporting Information: Study Protocol
Time Frame: Data and materials will be shared concurrent with publication and will be available indefinitely on the Open Science Framework.
Access Criteria: Anyone who wishes to access the data will be able to do so